CLINICAL TRIAL: NCT01088321
Title: Safety of Disease Modifying Antirheumatic Drug (DMARD) and Biologic Treatment of Rheumatoid Arthritis
Brief Title: Safety Study of Abatacept to Treat Rheumatoid Arthritis (A)
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IM101-045A
Record Dates: First submitted 2010-03-12; First posted 2010-03-17 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Patients initiating abatacept
- Patients initiating other biologic disease-modifying drugs
- Pts initiate non-biologic disease-modify anti-rheumatic drugs

SUMMARY:
The purpose of this study is to compare the incidence rates of infection among patients with rheumatoid arthritis who are treated with abatacept and those who are treated with other anti-rheumatic medications

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of rheumatoid arthritis
* Claims indicating infusion, injection, or dispensing of abatacept, a DMARD, or a BDM
* Age 18 years or older at the time of drug initiation
* Enrollment in the health plan at least 6 continuous months leading up to the time of study drug initiation

Exclusion Criteria:

* Below 18 years of age at the time of BDM or DMARD initiation
* Lacking six months of continuous enrollment prior to the initiation of one of the study drugs

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: United Healthcare
Sampling Method: Non-Probability Sample
Enrollment: 81332 (Actual)
Dates: Start 2005-03; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Infections, specifically hospitalized infection, hospitalized pneumonia, hospitalized and/or IV treated pneumonia, tuberculosis, herpes zoster, and opportunistic infection | Every four months throughout the study

SECONDARY OUTCOMES:
Anaphylactic reactions | Every four months throughout the study
Multiple sclerosis, lupus, and psoriasis | Every four months throughout the study
Concomitant biologic use | Every four months throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb